CLINICAL TRIAL: NCT03271177
Title: The PRAGMATIC Study:A Prospective Randomized Clinical Trial Comparing Radial Artery Intimal Hyperplasia Resulting From a 7F Sheathless Guide (Mach 1TM) vs. a 6F Transradial Sheath/Guide Combination in Coronary Intervention
Brief Title: Ultrasound Comparison of Radial Artery Hyperplasia After Use of a 7F Sheathless Guide vs. 6F Sheath/Guide Combination
Acronym: PRAGMATIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tallahassee Research Institute, Inc. (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-04
Record Dates: First submitted 2017-08-23; First posted 2017-09-01 (Actual); Last update posted 2017-09-01 (Actual); Status verified 2017-08

CONDITIONS: Coronary Artery Disease
Keywords: transradial percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 7F Sheathless Guide Catheter (Experimental): Patients in this arm will undergo their percutaneous coronary intervention using a 7F Sheathless guide catheter
  Interventions: Device: 7F sheathless Guide Catheter
- 6F Sheath/Guide Catheter Combination (Placebo Comparator): Patients in this arm will undergo their percutaneous coronary intervention using a 6F Sheath/guide combination
  Interventions: Device: 6F Sheath/Guide Catheter Combination

INTERVENTIONS:
Device: 7F sheathless Guide Catheter — Transradial PCI will be performed with a 7F sheathless Guide Catheter
  Arms: 7F Sheathless Guide Catheter
Device: 6F Sheath/Guide Catheter Combination — Transradial PCI will be performed with a 6F Sheath/Guide Catheter Combination
  Arms: 6F Sheath/Guide Catheter Combination

SUMMARY:
The purpose of this study is to determine if the routine use of a sheathless 7F guide catheter for transradial percutaneous coronary intervention (TR PCI) is non-inferior to a 6F sheath/guide combination with regards to radial artery injury (radial artery intimal-medial-adventitial thickening). To evaluate the radial artery, ultrahigh resolution ultrasonography (55 mHz) will be used to accurately quantify radial artery intimal-medial-adventitial thickness (IMT) at baseline and 90 days. A non-inferiority analysis will be performed to compare the degree of radial artery IMT at 90 days between the 7F sheathless guide approach and the 6F sheath/guide combination.

DETAILED DESCRIPTION:
The purpose of the PRAGMATIC study (A Prospective Randomized Trial comparing Radial Artery Intimal Hyperplasia resulting from a 7F Transradial Sheathless Guide [Mach 1] vs. a 6F Transradial Sheath/Guide Combination in Coronary Intervention) is 3 fold: (1) to determine if the routine use of a simple inexpensive "home-made" 7F sheathless guide catheter approach for TRA-PCI was associated with comparable degrees of radial artery access site injury and intimal-medial thickening (IMT) as the routine use of a 6F standard sheath/guide catheter combination; (2) to determine if the 7F sheathless approach was associated with comparable procedural success rates, procedure times, number of guides and crossover rates to a femoral approach compared to a 6F sheath/guide combination; and (3) to use ultrahigh resolution ultrasound to characterize the degree of RA injury and intimal-medial hyperplasia (IMT) that routinely occurs following transradial percutaneous coronary intervention.

Materials and Methods

Subjects and Study Design The study enrolled 41 consecutive patients undergoing elective non-emergent TRA-PCI at Tallahassee Memorial Hospital (TMH) from June 2016 to December 2016. The study protocol was approved by the TMH institutional review board. Informed consent was obtained prior to diagnostic coronary arteriography. Patients aged 21 years and over who were undergoing planned non-emergent PCI and willing to undergo a 24 hour and 90day post PCI RA ultrasound were eligible. Patients were excluded if they had undergone a prior ipsilateral TRA heart catheterization or PCI. There were no angiographic exclusions. Baseline clinical, demographic and angiographic characteristics were collected prospectively. Patients were randomly assigned to undergo TRA-PCI using a 7F sheathless Mach 1TM (Boston Scientific, Marlborough, MA) guide catheter or using our catheterization lab's standard 6F CordisTM (Johnson and Johnson, Inc.) sheath/6F Mach1TM guide combination. In order to minimize radial artery size bias, randomization was stratified according to patient sex. PCI with a drug-eluting stent was performed according to routine local practice and physician discretion. Patients were preferentially treated with a SYNERGYTM (Boston Scientific, Marlborough, MA) drug-eluting stent as the primary stent choice, however, other stents were allowed according to physician discretion.

All patients received dual antiplatelet therapy (DAPT) prior to TRA-PCI with an oral aspirin (325 mg) and a p2Y12 platelet inhibitor (either 600mg clopidogrel or 180mg ticagrelor) bolus. Intravenous heparin was administered to achieve an activated clotting time (ACT) of at least 300 seconds. Immediately following TRA-PCI, the sheath and/or guide was removed and RA hemostasis was achieved using a standardized and previously validated patent hemostasis protocol that incorporates the Terumo TR Band Radial Compression DeviceTM.

The technique used for the sheathless introduction of the 7F guide catheter was as follows: following diagnostic coronary angiography, a 6F 100 cm length multipurpose catheter (MP) was telescoped through the inner lumen of a 90 cm 7F Mach 1TM guide catheter. The MP was then used as an obturator to facilitate insertion of the 7F guide through the skin and into the RA arteriotomy site over a 0.035 J wire. Only after the 7F guide/6F MP combination was introduced into the RA and advanced together back to the aortic root, were the inner 6F MP catheter and 0.035 wire removed and the 7F guide engaged into the coronary ostium for TRA-PCI.

Ultrahigh Resolution Ultrasound Assessment Using the FDA approved FUJIFILM VisualSonics 55 mHz probe and previously established methods,16,17 ultrahigh resolution duplex ultrasound of the RA access site was performed at 24 hours (pre-discharge) and 90 days post TRA-PCI. This technique has been well validated as a means to accurately depict and quantify the individual layers of muscular and elastic arteries. To prevent RA vasospasm, sublingual nitroglycerin (0.4 mg) was administered within 3-5 minutes prior to performing the ultrasound studies. M-mode, 2-dimensional and color doppler images were obtained. The RA diameter was recorded and then the individual borders of the layers of the artery delineated with M-mode ultrasound. To determine the mean IMT, we started off with the center of the probe centered over the RA puncture site and recorded the thickest IMT measurements noted just proximal to the site, at the center of the site (center of probe) and just distal to the site. We then repositioned the probe more proximally, placing its distal leading edge at the puncture site and obtained another proximal and mid probe measurement of IMT. The final recorded IMT was the average of these 5 measurements. Using this technique, we ensured sampling over an adequate length of the RA proximal to, at and slightly distal to the point of arterial access.

The RA access site was also assessed for other signs of trauma, including small focal intimal tears, frank arterial dissections, pseudoaneurysms, arteriovenous fistulae, and vessel occlusion. Given high resolution imaging, we were forced to distinguish between limited focal intimal tears that were now easily visualized and simply a result of access site entry from more frank dissections. For this, we defined a limited access site intimal tear (LASIT) as a focal tear in the intima that was restricted to and not beyond the access site itself which did not encroach on the lumen or cause any flow abnormality. Tears or dissections beyond this were deemed true dissections. All studies and measurements were performed by 2 experienced vascular technicians who were blinded to treatment allocation with additional independent review by a reading physician who was also blinded to treatment allocation.

Other Clinical Endpoints Assessed:

Procedural success rates (successful implantation of the stent with residual stenosis of < 30% and no other complications), fluoroscopy time, the number of guide catheters used, and the frequency of cross-over from radial access to femoral access were also recorded. Routine clinical and interventional outcomes, including PCI success, in-hospital death, MI, coronary dissection, urgent revascularization were also prospectively collected. Ultrahigh frequency ultrasound parameters related

Statistical Analysis For comparisons between groups, two-sided Student t-tests were used for continuous variables and chi-square or Fisher exact tests for discrete variables. The primary outcome of the study was a comparison of radial artery IMT thickness at 90 days between the 7F sheathless guide catheter group and the standard 6F sheath/guide combination group. The primary statistical analysis was based on a non-inferiority analysis and an intention to treat design. The null hypothesis was that the 7F sheathless Mach 1TM guide would be associated with at least a 0.08mm increase in IMT at 90 days compared with the 6F sheath/guide combination. A non-inferiority margin of 0.08 mm was selected as this represented a relatively small change compared to baseline IMT and RA diameter (~25% of baseline IMT and only ~3% of RA diameter). It was therefore deemed unlikely that this small difference would be clinically significant. Based on our own pilot data and a prior study, a standard deviation of 0.08mm was assumed for IMT measurements. Assuming a one-sided 95% confidence interval, at least 36 evaluated patients (~18 per group) were needed to have 90% power to detect if the lower limit of the one-sided confidence interval lies above the 0.08 limit. If the 95% confidence interval lies below this 0.08mm boundary, then the null hypothesis was to be rejected and non-inferiority declared. Superiority testing was also applied using a p<0.05 for a level of significance for intergroup comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above with coronary artery disease
* Scheduled for transradial PCI

Exclusion Criteria:

* Has had prior transradial access for heart catheterization or PCI in same radial artery as planned access site
* Not willing to undergo follow-up ultrasound examinations
* Acute ST elevation myocardial infarction or other emergent PCI
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-02-25 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-13 (Actual)

PRIMARY OUTCOMES:
Radial artery access site intimal-medial thickness (IMT) | 90-day
  The incidence of other vascular complications such as radial artery occlusion, pseudo-aneurysms, radial artery diameter, and radial artery dissections will also be assessed.

SECONDARY OUTCOMES:
Procedural Success Rate | up to 24 hours
  Procedural Success Rate (successful coronary stent implantation with < 30% residual stenosis and no other complications)
Major Adverse Cardiac Events (MACE) | from date of PCI until date of death, MI or urgent revascularization, whichever came first, assessed up to 72 hrs
  In-hospital MACE (death, MI, urgent revascularization)
Fluoroscopy Time | During PCI procedure (from beginning of procedure until end)
  Fluoroscopy Time
Number of Guide Catheters Used | During PCI procedure (from beginning of procedure until end)
  Number of Guide Catheters Used during the procedure
Frequency of Cross-over from Radial Access to Femoral Access | During PCI procedure (from beginning of procedure until end)
  Rate of Needing to Cross-over from Radial Access to Femoral Access

CONTACTS AND LOCATIONS:
Overall Officials: Wayne B Batchelor, MD, MHS, Principal Investigator — Tallahassee Research Institute

IPD SHARING:
Plan to Share IPD: No